CLINICAL TRIAL: NCT00647738
Title: Single Dose Crossover Comparative Bioavailability Study of Baclofen 20 mg Tablets in Healthy Male Volunteers / Fasting State
Brief Title: Comparative Bioavailability Study of Baclofen 20 mg Tablets in Healthy Male Volunteers / Fasting State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Collaborators: Genpharm ULC (Industry)
Responsible Party: Elliot Offman, Director, Biopharmaceutics, Genpharm ULC
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BCE-P3-022
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Baclofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Baclofen
- 2 (Active Comparator)
  Interventions: Drug: Baclofen

INTERVENTIONS:
Drug: Baclofen — Single-dose 20 mg immediate-release oral tablets
  Arms: 1
Drug: Baclofen — Single-dose 20 mg immediate-release oral tablet
  Other Names: Lioresal®
  Arms: 2

SUMMARY:
The objective of this study was to investigate the bioequivalence of Genpharm's baclofen tablets following a single, oral 20 mg (1 x 20 mg) dose compared to the Baclofen USP (Watson Laboratories Inc., USA) administered under fasting conditions. Twenty-seven (27) healthy, light-, non- or ex-smoking subjects of at least 18 a years of age were randomized, in this two-period, two-treatment crossover bioequivalence study conducted by Eric Sicard, M.D. at Algorithme Pharma Inc. Montreal, Canada.

Statistical analysis of the data reveals that 90% confidence intervals are within the acceptable bioequivalent range of 80% and 125% for the natural log transformed parameters AUCT, AUCI and Cmax. This study demonstrates that Genpharm's baclofen 20 mg tablets are bioequivalent to Baclofen USP 20 mg tablets (Watson Laboratories Inc., USA) administered under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria may be included in the study: Availability of subject for the entire study period and willingness to adhere to protocol requirements as evidenced by the informed consent form duly signed by the subject

Males aged from 18 to 55 years with a body mass index (BMI) greater than or equal to 19 and below 30; demographic data (sex, age, ethnic group, body weight, height and smoking habits) will be recorded and reported in the final report

Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance and must be recorded as such in the CRF (laboratory tests are presented in section 7.1.3)

Healthy according to the laboratory results and physical examination

Normal cardiovascular function according to ECG

Subjects should be light-, non- or ex-smokers

Exclusion Criteria:

Significant history of hypersensitivity to baclofen or any related products as well as severe hypersensitivity reactions (like angioedema) to any drugs

Presence or history of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects

Presence or history of significant cardiovascular, pulmonary, hematologic, neurologic, psychiatric, endocrine, immunologic or dermatologic disease

Presence or history of urologic disease

Presence or history of neuromuscular disease

Maintenance therapy with any drug, or significant history of drug dependency, alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic), or serious psychological disease

Any clinically significant illness in the previous 28 days before day 1 of this study

Use of enzyme-modifying drugs in the previous 28 days before day 1 of this study (all barbiturates, corticosteroids, phenylhydantoins, etc.)

Participation in another clinical trial in the previous 28 days before day 1 of this study

Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study

Positive urine screening of drugs of abuse (drug names are presented in section 7.1.4)

Positive results to HIV, HBsAg or anti-HCV tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2003-10; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma, Montreal, Quebec, Canada

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html